CLINICAL TRIAL: NCT00769522
Title: Phase III Trial of Combined Immunochemotherapy With Fludarabine, Cyclophosphamide and Rituximab (FCR) Versus Bendamustine and Rituximab (BR) in Patients With Previously Untreated Chronic Lymphocytic Leukaemia
Brief Title: FCR or BR in Patients With Previously Untreated B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Roche Pharma AG (Industry); Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL10; CDR0000616169 (Other: Clinical Data Repository); 2007-007587-21 (EudraCT Number)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Bendamustine Hydrochloride; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FCR (Experimental)
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine
- BR (Experimental)
  Interventions: Biological: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Biological: Rituximab — cycle 1: 375 mg/m² i.v., day 0, q28d
  cycle 2-6: 500 mg/m² i.v., day 1, q28d
  Other Names: Mabthera; Rituxan
Drug: Bendamustine — cycle 1-6: 90mg/m² i.v., day 1-2, q28d
  Other Names: Levact; Ribomustin; Treanda
  Arms: BR
Drug: Cyclophosphamide — cycle 1-6: 250 mg/m² i.v., days 1-3, q28d
  Other Names: Endoxan
  Arms: FCR
Drug: Fludarabine — cycle 1-6: 25 mg/m² i.v., days 1-3, q28d
  Other Names: Fludura
  Arms: FCR

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, cyclophosphamide, and bendamustine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving fludarabine and cyclophosphamide together with rituximab is more effective than giving bendamustine together with rituximab in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying fludarabine, cyclophosphamide, and rituximab to see how well they work compared with bendamustine and rituximab in treating patients with previously untreated B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the therapeutic efficacy of fludarabine phosphate, cyclophosphamide, and rituximab vs bendamustine hydrochloride and rituximab in patients with previously untreated B-cell chronic lymphocytic leukemia.
* To compare the incidence of major side effects (e.g., myelosuppression) associated with these regimens in these patients.
* To compare the rate of infections and secondary neoplasias in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to country and disease stage. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine phosphate IV and cyclophosphamide IV on days 1-3. Patients also receive rituximab IV on day 0 of course 1 and on day 1 of courses 2-6. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive bendamustine hydrochloride IV on days 1 and 2. Patients also receive rituximab as in arm I. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life questionnaires (EORTC-C30 and EURO-QOL) at baseline and then at 12, 24, 36, 48, and 60 months.

After completion of study therapy, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then once a year thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of B-cell chronic lymphocytic leukemia (CLL) meeting 1 of the following criteria:
* Binet stage C disease or stage B or A disease requiring treatment
* Binet stage B or A disease meeting ≥ 1 of the following:
* B-symptoms (e.g., night sweats, weight loss ≥ 10% within the past 6 months, fevers > 38°C or 100.4°F for ≥ 2 weeks without evidence of infection) or constitutional symptoms (e.g., fatigue)

  * Progressive lymphocytosis, defined as peripheral lymphocyte count > 5 x 10^9/L (i.e., > 50% increase over a 2-month period or doubling of peripheral blood lymphocyte count < 6 months)
  * Evidence of progressive marrow failure as manifested by the development/worsening of anemia and/or thrombocytopenia
  * Massive, progressive, or painful splenomegaly or hypersplenism
  * Massive lymph nodes or lymph node clusters (> 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy

    * No 17p deletion by FISH
    * No aggressive B-cell cancer, such as Richter syndrome

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 6 months
* Total bilirubin ≤ 2 times upper limit of normal (ULN) (unless directly attributable to CLL)
* AST and ALT ≤ 2 times ULN (unless directly attributable to CLL)
* Creatinine clearance ≥ 70 mL/min (creatinine clearance is to be calculated only in patients with serum creatinine ≥ 1.1 mg/dL)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* Hepatitis B and C negative
* HIV negative
* CIRS score > 6 or a single score of 4 for one organ category
* No active secondary malignancy requiring treatment, except basal cell carcinoma or malignant tumor curatively treated by surgery, or successfully treated secondary malignancies in complete remission > 5 years prior to enrollment
* No history of anaphylaxis following exposure to monoclonal antibodies
* No active bacterial, viral, or fungal infection
* No medical condition requiring prolonged use of oral corticosteroids (i.e., > 1 month)
* No cerebral dysfunction or legal incapacity
* No circumstance that would preclude completion of the study or the required follow-up

PRIOR CONCURRENT THERAPY:

* No prior CLL specific-chemotherapy, radiotherapy, and/or immunotherapy

  * Prednisolone administered immediately prior to initiation of study therapy allowed for very high lymphocyte counts
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2008-10-02 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate after 24 months | 2008-2015
  estimated time point when 198 needed events for the final analysis(PD or deaths) have occured.

SECONDARY OUTCOMES:
Minimal residual disease, complete response rates, and partial response rates | 2008-2015
  done within the final analysis
Duration of remission | 2008-2015
  done within the final analysis
Event-free survival | 2008-2015
  done within the final analysis
Overall survival | 2008-2015
  done within the final analysis
Overall response rate | 2008-2015
  done within the final analysis
Response rates in and survival times in biological subgroups | 2008-2015
  done within the final analysis
Toxicity rates | 2008-2015
  done within the final analysis
Quality of life | 2008-2015
  done within the final analysis
Standard safety analysis | 2008-2015
  done within the final analysis

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Eichhorst, MD, Principal Investigator — Medizinische Universitaetsklinik I at the University of Cologne
Locations (1):
- Medizinische Universitaetsklinik I at the University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz DM, Esfahani MS, Scherer F, Soo J, Jin MC, Liu CL, Newman AM, Duhrsen U, Huttmann A, Casasnovas O, Westin JR, Ritgen M, Bottcher S, Langerak AW, Roschewski M, Wilson WH, Gaidano G, Rossi D, Bahlo J, Hallek M, Tibshirani R, Diehn M, Alizadeh AA. Dynamic Risk Profiling Using Serial Tumor Biomarkers for Personalized Outcome Prediction. Cell. 2019 Jul 25;178(3):699-713.e19. doi: 10.1016/j.cell.2019.06.011. Epub 2019 Jul 4. PMID 31280963
- [Background] Dimier N, Delmar P, Ward C, Morariu-Zamfir R, Fingerle-Rowson G, Bahlo J, Fischer K, Eichhorst B, Goede V, van Dongen JJM, Ritgen M, Bottcher S, Langerak AW, Kneba M, Hallek M. A model for predicting effect of treatment on progression-free survival using MRD as a surrogate end point in CLL. Blood. 2018 Mar 1;131(9):955-962. doi: 10.1182/blood-2017-06-792333. Epub 2017 Dec 18. PMID 29255066
- [Background] Kutsch N, Robrecht S, Fink A, Lange E, Weide R, Kiehl MG, Sokler M, Schlag R, Vehling-Kaiser U, Kochling G, Ploger C, Gregor M, Plesner T, Clausen MR, Oschlies I, Ritgen M, Herling M, Fischer K, Dohner H, Wendtner CM, Kreuzer KA, Stilgenbauer S, Hallek M, Bottcher S, Klapper W, Eichhorst B. The role of trephine bone marrow biopsies in the era of measurable residual disease-Results from the CLL10 trial of the German CLL Study Group (GCLLSG). Hemasphere. 2024 Jul 24;8(7):e126. doi: 10.1002/hem3.126. eCollection 2024 Jul. No abstract available. PMID 39050548
- [Background] Eichhorst B, Fink AM, Bahlo J, Busch R, Kovacs G, Maurer C, Lange E, Koppler H, Kiehl M, Sokler M, Schlag R, Vehling-Kaiser U, Kochling G, Ploger C, Gregor M, Plesner T, Trneny M, Fischer K, Dohner H, Kneba M, Wendtner CM, Klapper W, Kreuzer KA, Stilgenbauer S, Bottcher S, Hallek M; international group of investigators; German CLL Study Group (GCLLSG). First-line chemoimmunotherapy with bendamustine and rituximab versus fludarabine, cyclophosphamide, and rituximab in patients with advanced chronic lymphocytic leukaemia (CLL10): an international, open-label, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2016 Jul;17(7):928-942. doi: 10.1016/S1470-2045(16)30051-1. Epub 2016 May 20. PMID 27216274
- [Background] Kovacs G, Robrecht S, Fink AM, Bahlo J, Cramer P, von Tresckow J, Maurer C, Langerbeins P, Fingerle-Rowson G, Ritgen M, Kneba M, Dohner H, Stilgenbauer S, Klapper W, Wendtner CM, Fischer K, Hallek M, Eichhorst B, Bottcher S. Minimal Residual Disease Assessment Improves Prediction of Outcome in Patients With Chronic Lymphocytic Leukemia (CLL) Who Achieve Partial Response: Comprehensive Analysis of Two Phase III Studies of the German CLL Study Group. J Clin Oncol. 2016 Nov 1;34(31):3758-3765. doi: 10.1200/JCO.2016.67.1305. PMID 27573660
- [Background] Al-Sawaf O, Robrecht S, Bahlo J, Fink AM, Cramer P, von Tresckow J, Maurer C, Bergmann M, Seiler T, Lange E, Kneba M, Stilgenbauer S, Dohner H, Kiehl MG, Jager U, Wendtner CM, Fischer K, Goede V, Hallek M, Eichhorst B, Hopfinger G. Impact of gender on outcome after chemoimmunotherapy in patients with chronic lymphocytic leukemia: a meta-analysis by the German CLL study group. Leukemia. 2017 Oct;31(10):2251-2253. doi: 10.1038/leu.2017.221. Epub 2017 Jul 12. No abstract available. PMID 28745332
- See also: Click here for more information about this study: CLL10 (German CLL Study Group) — https://www.dcllsg.com/cll10/